CLINICAL TRIAL: NCT00856843
Title: BLI800-303: An Efficacy Evaluation of 2 Different Bowel Cleansing Preparations in Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Associate Director, Clinical Research, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI800-303
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-10

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyethylene glycol 3350 based bowel preparation (Active Comparator): Polyethylene glycol 3350 based bowel preparation
  Interventions: Drug: Polyethylene glycol 3350 based bowel preparation
- BLI800 (Experimental): BLI800
  Interventions: Drug: BLI800

INTERVENTIONS:
Drug: BLI800 — Solution for oral administration prior to colonoscopy
  Arms: BLI800
Drug: Polyethylene glycol 3350 based bowel preparation — Solution for oral administration prior to colonoscopy
  Arms: Polyethylene glycol 3350 based bowel preparation

SUMMARY:
To evaluate the safety and efficacy of BLI800 vs an FDA approved bowel preparation before colonoscopic examination in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
2. At least 18 years of age
3. Otherwise in good health, as determined by physical exam and medical history
4. If female, and of child-bearing potential, is using an acceptable form of birth control
5. Negative urine pregnancy test at screening, if applicable
6. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

1. Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
2. Subjects who had previous gastrointestinal surgeries.
3. Subjects with known or suspected electrolyte abnormalities such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalemia, hypocalcemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
4. Subjects with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
5. Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
6. Subjects undergoing colonoscopy for foreign body removal and decompression.
7. Subjects who are pregnant or lactating, or intending to become pregnant during the study.
8. Subjects of childbearing potential who refuse a pregnancy test.
9. Subjects allergic to any preparation components
10. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
11. Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (5):
- United States (5):
  - University of South Alabama, Mobile, Alabama
  - Jupiter Research, Jupiter, Florida
  - Miami Research Associates, Miami, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Long Island GI Research Group, Great Neck, New York

REFERENCES:
- [Derived] Rex DK, Di Palma JA, Rodriguez R, McGowan J, Cleveland M. A randomized clinical study comparing reduced-volume oral sulfate solution with standard 4-liter sulfate-free electrolyte lavage solution as preparation for colonoscopy. Gastrointest Endosc. 2010 Aug;72(2):328-36. doi: 10.1016/j.gie.2010.03.1054. Epub 2010 Jun 19. PMID 20646695

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyethylene Glycol 3350 Based Bowel Preparation: Active control - oral solution, 1 administration
- BLI800: Investigational prep - oral solution, 1 administration
Period: Overall Study
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Started | 68 | 68
Completed | 66 | 63
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800 | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 50 | 103
  >=65 years | 15 | 18 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.0) | 57.7 (10.8) | 57.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 37 | 32 | 69
Region of Enrollment [Number; unit: participants]
  United States | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage of Patients With Successful Preparations Based on a 4 Point Scale
Description: Blinded colonoscopists rated cleansing quality as either Excellent, Good, Fair or Poor. Scores of Excellent or Good were considered Successful preparations.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants | 89.6 | 98.4
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.038, Chi-squared; Difference in success rates = 8.8, 95% CI 2-sided [0.9 to 16.8]

2. Secondary Outcome: Assessment of Residual Stool - Cecum
Description: The blinded colonoscopist rated residual stool in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 67 | 91
  Small | 22 | 9
  Moderate | 5 | 0
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.010, Chi-squared

3. Secondary Outcome: Assessment of Residual Stool - Ascending Colon
Description: The blinded colonoscopist rated residual stool in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 69 | 91
  Small | 24 | 9
  Moderate | 2 | 0
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.020, Chi-squared

4. Secondary Outcome: Assessment of Residual Stool - Transverse Colon
Description: The blinded colonoscopist rated residual stool in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 82 | 92
  Small | 9 | 8
  Moderate | 2 | 0
  Excess | 2 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.644, Chi-squared

5. Secondary Outcome: Assessment of Residual Stool - Descending Colon
Description: The blinded colonoscopist rated residual stool in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 84 | 92
  Small | 9 | 8
  Moderate | 2 | 0
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.763, Chi-squared

6. Secondary Outcome: Assessment of Residual Stool - Sigmoid Colon/Rectum
Description: The blinded colonoscopist rated residual stool in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 81 | 94
  Small | 10 | 5
  Moderate | 5 | 1
  Excess | 3 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.173, Chi-squared

7. Secondary Outcome: Assessment of Residual Fluid - Cecum
Description: The blinded colonoscopist rated residual fluid in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 15 | 43
  Small | 63 | 44
  Moderate | 15 | 13
  Excess | 2 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.004, Chi-squared

8. Secondary Outcome: Assessment of Residual Fluid - Ascending Colon
Description: The blinded colonoscopist rated residual fluid in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 36 | 64
  Small | 43 | 36
  Moderate | 15 | 0
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Assessment of Residual Fluid - Transverse Colon
Description: The blinded colonoscopist rated residual fluid in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 49 | 68
  Small | 30 | 32
  Moderate | 13 | 0
  Excess | 12 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.005, Chi-squared

10. Secondary Outcome: Assessment of Residual Fluid - Descending Colon
Description: The blinded colonoscopist rated residual fluid in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 39 | 67
  Small | 48 | 27
  Moderate | 8 | 6
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.013, Chi-squared

11. Secondary Outcome: Assessment of Residual Fluid - Sigmoid Colon/Rectum
Description: The blinded colonoscopist rated residual fluid in specific colon sections as Absent, Small, Moderate or Excess.
Time Frame: 2 days
Measure: Number; unit: percentage of participants
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
percentage of participants
  Absent | 48 | 64
  Small | 42 | 32
  Moderate | 8 | 5
  Excess | 0 | 0
Statistical Analysis 1: Comparison: Polyethylene Glycol 3350 Based Bowel Preparation vs BLI800; Test type: Superiority or Other; p = 0.283, Chi-squared

12. Secondary Outcome: Subject Symptom Scores
Description: Expected preparation related symptoms of Abdominal Cramping, Abdominal Bloating, Nausea and Overall discomfort were rated by each subject from 1 - 5 (1=none, 2=mild, 3=bothersome, 4=distressing, 5=severely distressing).
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
units on a scale
  Cramping | 1.21 (0.45) | 1.33 (0.60)
  Stomach bloating | 1.62 (0.84) | 1.33 (0.54)
  Nausea | 1.82 (1.08) | 1.54 (0.71)
  Overall discomfort | 1.77 (0.94) | 1.65 (0.70)

13. Secondary Outcome: Mean Change in Serum Chemistry (mg/dL)
Description: Mean changes from Baseline to Post-preparation for the following analytes will be compared between treatment groups: blood urea nitrogen, calcium, creatinine, phosphorus. Baseline lab samples were allowed to be drawn within 15 days of the post-preparation (Visit 2) lab draw.
Time Frame: up to 15 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
mg/dL
  Blood Urea Nitrogen | -3.95 (3.3) | -3.78 (3.5)
  Calcium | -0.24 (0.45) | -0.19 (0.49)
  Creatinine | 0.02 (0.09) | 0.01 (0.1)
  Phosphorus | -0.10 (0.53) | -0.18 (0.99)

14. Secondary Outcome: Mean Change in Serum Chemistry (mEq/L)
Description: Mean changes from Baseline to Post-preparation for the following analytes will be compared between treatment groups: bicarbonate, chloride, magnesium, potassium, sodium. Baseline lab samples were allowed to be drawn within 15 days of the post-preparation (Visit 2) lab draw.
Time Frame: up to 15 days
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Number analyzed (Participants) | 67 | 63
mEq/L
  Bicarbonate | -0.81 (2.0) | -1.76 (2.0)
  Chloride | 0.66 (2.4) | -0.37 (2.5)
  Magnesium | -0.04 (0.11) | 0.04 (0.13)
  Potassium | -0.16 (0.47) | 0.03 (0.64)
  Sodium | 0.36 (2.2) | 0.09 (2.4)

ADVERSE EVENTS:
Arm/Group | Polyethylene Glycol 3350 Based Bowel Preparation | BLI800
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/63
Other Adverse Events (participants affected / at risk) | 6/67 | 1/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyethylene Glycol 3350 Based Bowel Preparation (N=67) | BLI800 (N=63)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyethylene Glycol 3350 Based Bowel Preparation (N=67) | BLI800 (N=63)
nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
As prespecified in the study protocol, expected prep related side effects (nausea, vomiting, cramping, bloating and overall discomfort) were only documented as AEs if patients rated them severely distressing on the study questionnaire.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 360 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo.